CLINICAL TRIAL: NCT04775381
Title: Study of Total Post-thyroidectomy Hypocalcemia After Preoperative Cholecalciferol Supplementation
Brief Title: Total Post-thyroidectomy Hypocalcemia After Preoperative Cholecalciferol Supplementation
Acronym: CAVITHY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHRD 2115; 2018-000526-64 (EudraCT Number)
Record Dates: First submitted 2021-02-19; First posted 2021-03-01 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Hypocalcemia
Keywords: Total thyroidectomy; hypocalcemia; cholecalciferol supplementation
MeSH Terms: conditions — Hypocalcemia | interventions — Vitamin D; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): During preoperative visit (Month -2) patients will receive a cholecalciferol supplementation added to a fruit juice.
  Interventions: Drug: Vitamin D
- Fruit juice (No Intervention): During preoperative visit (Month -2) patients will receive only fruit juice.

INTERVENTIONS:
Drug: Vitamin D — Patients will receive a cholecalciferol supplementation added to a fruit juice.
  Other Names: Treatment
  Arms: Vitamin D

SUMMARY:
This prospective study evalue the inflence of pre operative vit D3 administration on post operative hypocalcemia in patients undergoing Total thyroidectomy

DETAILED DESCRIPTION:
Thyroidectomy is a frequent procedure. This surgery is well known but not devoid of risks. The most common postoperative complication is transitory hypocalcemia. Some studies have reported that preoperative vitamin D deficiency (VDD) is a risk factor for hypocalcemia after total thyroidectomy (TT) in patients with non toxic multinodular goiter or graves's disease. Although the association between VVD and postoperative hypocalcemia in thyroid cancer patients undergoing TT plus central compartment neck dissection (CCND) remains unclear. This prospective study evalue the inflence of pre operative vit D3 administration on post operative hypocalcemia in patients undergoing TT.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient shall be operated on for a total thyroidectomy in one time for any indication
* Written informed consent (IC) obtained
* Patients with affiliation to the social security system

Exclusion Criteria:

• Medical history of : Thyroid or parathyroid surgery Hyperparathyroidism Granulomatosis flare-up

* Hypocalcemia, hypercalcemia/ hypercalciuria, or symptom of Hypocalcemia, hypercalcemia/ hypercalciuria, not due to thyroid pathologies
* Chronic kidney disease grade ≥4
* Severe liver failure
* 25OHD supplementation within last 3 months before surgery
* Malabsorption syndrome
* Known hypersensitivity to vitamin D
* Medical history of calcic lithiasis
* Pregnant women
* Vulnerable populations (guardianship or trusteeship)
* Allergies to one of the components of the fruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effect of pre-operative cholecalciferol supplementation on the occurrence of post-operative hypocalcemia after total thyroidectomy | At Day 15 after surgery
  Measure of the occurrence of serum and / or clinical hypocalcemia.
  Serum hypocalcemia is defined by a level of calcemia, corrected for albuminemia, of less than 2.00 mmol / L.
  Clinical hypocalcemia is defined by the appearance of one of the following signs: sign of Chvostek, sign of Trousseau, paresthesias of the extremities and perioral between surgery and day 15

SECONDARY OUTCOMES:
Comparison of clinical course in both Arm | At 3 month
  Clinical course will be measured, for several items, and compared between both groups to see if a significant difference is observed.
  Items, considered for comparison, are listed below :
  * Initial hospital stay (number of days),
  * number of readmission,
  * adverse event (number)
Comparison of severity of hypocalcemia in both arm | At Day 1, Day 2 and Day 15
  The severity of hypocalcemia will be measured in both arm, to see if a significant difference is observed, with items listed below :
  * Calcemia, corrected for albuminemia, of less than 1.90 mmol / L
  * the use of calcium gluconate IV in the first 15 post-operative days)
  * duration of hypocalcemia's symptoms in the first 15 days postoperative
Comparison of the effect of supplementation on vitamin D deficiency in both arm | At Day 0
  Comparison between measured initial value of 25OHD at the inclusion visit to the measured value of 25OHD on the day of the operation in both groups.
Comparison of parathyroid activity in both arm | At Day 0 (= Surgery), at Hour 4 post-surgery, Day 2 and Day 15
  Parathyroid activity will be evaluated in both group by measuring parathormone (PTH).
  Hypoparathyroidism being defined by PTH < 15 ng / L.
Assessment of the prevalence of definitive hypocalcemia | At Day 15
  Collect of the definitive hypocalcemia's numbers in each group
Assessment of the effect of vitamin D supplementation on the occurrence of hypocalcemia in risk groups: hyperthyroidism, cancer, dissection associated with thyroidectomy | At Day 15
  Collect of the number of adverse events and serum calcium levels for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Dr Khaled AL TABAA, Principal Investigator — Hôpital NOVO
Locations (6):
- France (6):
  - Department of General, Digestive and Endocrine Surgery, Auxerre
  - Department of ENT and maxillofacial surgery, Corbeil-Essonnes
  - Department of Head and Neck Surgery and ENT, La Roche-sur-Yon
  - Hospital Lariboisière, Paris X, Paris
  - Hospital Poissy/Saint-Germain, Poissy
  - Hospital René Dubos,, Pontoise